CLINICAL TRIAL: NCT05664373
Title: The Use of Coronary Displaced Flap and Deepithelialized Free Graft in the Treatment of Multiple Adjacent Gingival Recessions - A Randomized Controlled Clinical Study
Brief Title: The Use of Coronary Displaced Flap and Deepithelialized Free Graft in the Treatment of Multiple Gingival Recessions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Natasa Nikolic Jakoba, Associate Professor, University of Belgrade
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EA 36/17
Record Dates: First submitted 2022-12-01; First posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Gingival Recession Generalized Moderate
Keywords: gingival recession; deepithelialized free gingival graft; coronally advanced flap; epithelial remnants
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- extraoraly de-epithelialized free gingival graft in combination with CAF (Active Comparator): Epithelium will be removed after harvesting the graft by using the blade. By using the blade the epithelium will be separated from the connective tissue.
  Interventions: Procedure: Coronally advanced flap and deepithelized free gingival graft
- intraoraly de-epithelialized free gingival graft in combination with CAF (Experimental): The epithelium will be removed prior to harvesting the graft from the palate. By using a diamond bur the epithelium will be removed until the connective tissue is exposed on the whole area of the intended graft size. Thereafter, the graft will be harvested.
  Interventions: Procedure: Coronally advanced flap and deepithelized free gingival graft

INTERVENTIONS:
Procedure: Coronally advanced flap and deepithelized free gingival graft — Free gingival grafts, de-epithelialized intraoraly or extraoraly in combination with coronally advanced flap will be used in the treatment of multiple gingival recessions.

SUMMARY:
Successful treatment of multiple gingival recessions (MRG) is a major challenge in periodontal plastic surgery due to complicated predisposing anatomical features of the surrounding tissues, such as a thin gingival phenotype or a limited zone of keratinized gingiva, variations in the depth and width of adjacent gingival recessions, shallow vestibulum and coronally inserted frenums and/or plica.The application of coronary advanced flap (CAF) or tunnel technique (TUN) with connective tissue graft (CTG) gives the best results in the therapy of MRG The application of connective tissue grafts in combination with various surgical techniques is accepted as the "gold standard" in GR therapy. A limitation in the application of CTG is the limited region of the donor site, especially in cases where a larger dimension of the CTG is required, or if the thickness of the hard palate tissue is inadequate. Techniques for obtaining subepithelial CTG (S-CTG), whether it is the trap-door technique or the single incision technique, are often associated with postoperative pain and discomfort, as well as necrosis/dehiscence of the palatal flap at the donor site.

In order to overcome these limitations and obtain a firmer and more uniform CTG, especially when the thickness of the palatal tissue is inadequate (≤2.5 mm) and when a large dimension of the graft in the apico-coronary or mesio-distal direction is required, deepithelialization of the free gingival graft has been proposed (D-FGG). D-FGG has also been shown to be less prone to postoperative contraction, as it consists predominantly of collagen-rich connective tissue from the lamina propria, while adipose/glandular tissue is minimally represented. FGG can be deepithelialized intraorally with a diamond bur or diode laser, or extraorally with a scalpel. Despite all the biological advantages of D-FGG, there is scarce evidence in the literature about its histological characteristics after intraoral and extraoral deepithelialization, as well as the clinical outcomes of grafts thus obtained in combination with CAF in the treatment of MGR. Therefore, this aims of the study are to investigate the clinical efficacy and postoperative patient morbidity using D-FGG and modified CAF in the treatment of MGR, as well as to evaluate the histological characteristics of grafts obtained using two different deepithelialization techniques.

DETAILED DESCRIPTION:
This study would be a single-centre, randomized clinical trial (RCT) and would be structured according to the CONSORT statement (http://vvv.consort-statement.org/).

The study would include 50 systemically healthy patients who came to the Clinic for Periodontology and Oral Medicine, School of Dental Medicine, University of Belgrade for the treatment of multiple gingival recessions, and who meet the inclusion criteria.

STUDY DESIGN The study will include patients who voluntarily gave and signed their consent to participate in the research based on written and oral information about the type, duration and expected outcome of the research (document attached).

Split mouth design will be applied in the study. Both sides of the same jaw will be treated using CAF and D-FGG. Immediately before the surgery, using computerized randomization tables,the method of de-epithelialization of the graft will be determined. The contralateral side will be treated no earlier than two months after the first surgical procedure, and FGG will be de-epithelialized using a technique that was not used in the previous intervention.

Clinical examination and initial therapy

After filling out the anamnestic sheet and signing the consent to participate in the study, the patient will undergo a periodontal examination. In order to verify the periodontal status and the level of oral hygiene, the following clinical parameters will be recorded:

* Periodontal probing depth (PPD)
* Clinical attachment level (CAL)
* Bleeding on probing (BOP)
* Plaque Index (PI) Clinical parameters will be recorded in six reference points (vestibulomesial, vestibulomedial, vestibulodistal, oromesial, oromedial, orodistal) on all present teeth (except third molars) using a periodontal probe (PCPUNC-15; HU-Friedy , Chicago, IL, USA). All measurements will be rounded to the nearest 0.5 mm and will be performed by a pre-calibrated dentist.

The following parameters will be measured on teeth with gingival recessions, at the mid-buccal point of the treated tooth:

* Recession depth (RD) - measured distance from the gingival margin to the CEJ.
* Recession width (RW) - horizontal dimension of gingival recession at the level of CEJ.
* Keratinized tissue width (KTW) - measured distance from the gingival margin to the mucogingival line (MGL), where the location of the MGL will be determined by the functional method
* Gingival thickness (GT) - will be measured in the middle of the buccal surface of the tooth, 1 mm apical from the bottom of the gingival sulcus, using an endodontic needle (K files, 10, FKG, Swiss Endo)

Clinical measurements will be recorded at the beginning of the study and 3, 6 and 12 months, 5 and 10 years after surgical therapy.

In the first visit, after anamnesis and clinical examination, patients will rinse their mouths with 15 ml of 0.12% chlorhexidine solution for 1 min (Curasept ADS 212, Curasept S.p.A. Saronno (VA), Italy), and then supra- and subgingival plaque and calculus will be removed using mechanical instruments (MiniPiezon, EMS Electro Medical Systems, Switzerland). After that, patients will be trained on proper maintenance of oral hygiene. Surgical therapy of gingival recession will be scheduled in case PI and BOP are <15%.

Surgical procedure All surgical procedures will be performed by the same surgeon (NNJ). After administration of local anesthesia, exposed root surfaces will be treated with Gracie's curettes (Hu-Friedy). The modified CAF will be formed in the region of the teeth behind the recessions and will include at least one more tooth mesial and distal to the tooth with gingival recession.

Oblique incisions in the area of the interdental papillae will prepare a half-thickness flap in order to form the so-called surgical papillae. These incisions will be joined by intrasulcular incisions, and then a full-thickness flap will be elevated in the area of the exposed roots by blunt dissection. Apicallly from the mucogingival line, in order to enable flap mobilization in the coronary direction, two incisions will be made: one to cut the periosteum, and the other to cut the muscles underneath mucosa. After that, the anatomical papillae will be deepithelialized. The D-FGG will be fixed at the recipient site with single sutures (5.0, Surgicryl Monofilament Polydioxanone, SMI AG, St. Vith Belgium), and then the flap will be sutured 1-2 mm more coronal than the CEJ with sling sutures (6.0, Polypropylene Blue, SMI AG).

In both groups, D-FGG will be taken in the region from the distal surface of the maxillary canine to the distal surface of the maxillary first/second molar. Intraoral deepithelialization of FGG will be performed using a 2.3 mm diameter diamond bur (801G/023, EMS, Aldrich Co.) with continuous application of saline (ID group), while the second group of grafts will be deepithelialized extraorally using a scalpel N°15C (Swann-Morton). to achieve an optimal thickness of 1-1.5 mm (ED group).

In both groups, for the purpose of better hemostasis and protection of the donor site from external influences, a gelatin sponge (Cutanplast©) will be placed on the hard palate in the wound area and fixed with crossed mattress sutures (5-0 silk sutures, Dogsan sutures, Trabzon, Turkey).

Immediately after separating the graft from the donor site, the thickness, length (mesial-distal dimension) and width (apical-coronal dimension) of the graft will be measured with a digital caliper (Alpha Tools Digital Caliper) with a resolution of 0.05. In the ED group, the thickness of the graft will be measured before and after deepithelialization. For histological analysis in both groups of grafts, they will take the most distal part of the graft, 2 mm wide, which will include the coronary and apical part of the graft.

The duration of graft deepithelialization in each group, as well as the total duration of surgical intervention will be recorded.

Post-surgical protocol All patients will be advised to avoid mechanical trauma, tooth brushing and flossing in the surgical regions during the postoperative two weeks until the sutures are removed. In order to achieve biofilm control, a 0.12% chlorhexidine-gluconate mouthwash solution will be prescribed 2 times a day for 1 min for 2 weeks.

Patients will be prescribed 600 mg of ibuprofen (Ibuprofen 600 mg, FAMARA S.A., Athens, Greece) immediately after surgery and one tablet 6 h after surgery. Also, they will be asked to record the additional intake of analgesics (number and dose) on a daily basis during the second week after surgery. After suture removal, 2 weeks after surgery, biofilm removal will begin with a soft toothbrush and rotary brushing technique. Two months after surgery, patients will be instructed to return to regular oral hygiene habits.

Pain intensity after the intervention will be evaluated with the help of the Visual Analogue Scale (VAS). By drawing a vertical line, on a scale whose value describes the degree of pain (0- complete absence of pain, and 10- the strongest possible pain), the patient will rate the pain he feels after the operation. The presence and intensity of pain will be recorded in the first 7 days, as well as 1, 3 and 6 months after surgery. On the first day, patients will assess discomfort 5 hours after surgery, as well as every morning between 8 a.m. and 10 a.m. for the next 7 days.

Also, an independent researcher will evaluate the aesthetic parameters of the surgically treated region 3, 6 and 12 months. 5 and 10 years after the intervention using the IRoot esthetic score.

HISTOLOGICAL ANALYSIS Histological analyzes will be performed by a senior oral pathologist (XX) who will not know by which procedure D-FGG was deepithelialized, in serial sections (5 sections for each sample). For the histological analysis of D-FGG samples, 2 mm long graft will be taken from the distal end of the graft and fixed in 10% neutral buffered formalin solution for 24 hours. After that, it will be rinsed with running water for 1 hour, then immersed in a 50% alcohol solution for 24 hours, after which it will be placed in a 70% alcohol solution and kept until further processing for histological analysis.

Samples were prepared on 5 mm thick histological sections and stained with hematoxylin-eosin (H&E) and Masson's trichrome stain. Assessment of the presence and abundance of epithelial remnants, inflammatory infiltrate and connective tissue cellularity will be performed on H&E sections.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years,
* Non-smokers or consumption of up to 10 cigarettes per day,
* no signs of gingival inflammation,
* Presence of at least two single-rooted teeth with type I gingival recession ≥2 mm deep on the buccal side on both sides of the jaw,
* Plaque index (PI) and gingival bleeding on provocation (BOP) <15% and probing depth (PPD) <3 mm,
* Absence of non-carious cervical lesions (NCL) and undetectable cemento-enamel junctionr (CEJ) at defect sites,
* No history of previous periodontal plastic surgery on the affected teeth.

Exclusion Criteria:

* Presence of carious lesions or restorations in the CEJ area,
* Use of medications that affect periodontal health and healing,
* Medical contraindications for periodontal surgical procedures,
* Pregnancy and breastfeeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-11-10 (Estimated); Study Completion 2034-12-10 (Estimated)

PRIMARY OUTCOMES:
the presence of the epithelial remnants in the D-FGG grafts | 2 years
  The presence of the epithelial remnants in the D-FGG grafts, wich were deepithelialized in different manner, will be histologically assessed

SECONDARY OUTCOMES:
Periodontal probing depth (PPD) | 10 years
  The distance from the gingival margin to the apical portion of the gingival sulcus using the periodontal probe.
postsurgery pain assessment | 2 months after surgery
  VAS will be used to assess postoperative patient morbidity parameters (postoperative pain, patient discomfort, tenderness, and bleeding) in relation to deepithelialization technique and graft size
Root esthetic score (RES) | 10 years
  assessment of esthetic parameters of the treated region after surgery
OHIP -14 | 1 year
  examination of the impact of surgical therapy of multiple recessions on the quality of life of patients
Gingival recession depth | 10 years
  measured at the mid-buccal aspect of the tooth from the CEJ to the most apical point of the GM.
Gingival recession width | 10 years
  measured at the mesiodistal direction of the gingival margin at the level of cementoenamel junction
Keratinized tissue width | 10 years
  measured as the distance between the gingival margin and the mucogingival junction
Clinical attachment level | 10 years
  measured at the mid-buccal aspect of the tooth from cementoenamel junction to the bottom of the sulcus
Gingival thickness | 10 years
  measured at the mid-buccal aspect of a treated tooth on the long axis, 3 mm apically from the gingival margin using K-file 25 ISO with a silicon marker driven perpendicularly to the gingival surface after application of local anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Natasa Nikolic Jakoba, DDS, PhD, Principal Investigator — School of Dental Medicine, University of Belgrade, Serbia
Locations (1):
- Natasa Nikolic Jakoba, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No